CLINICAL TRIAL: NCT06902584
Title: North American Comfilcon A Clinical Study
Status: Recruiting | Type: Observational
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: CV-24-19
Record Dates: First submitted 2025-03-11; First posted 2025-03-30 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Astigmatism; Presbyopia; Ametropia
MeSH Terms: conditions — Astigmatism; Presbyopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (5):
- comfilcon A Sphere Lens Wearers: Habitual comfilcon A Sphere Lens Wearers
  Interventions: Device: comfilcon A Sphere lens
- comfilcon A Toric Lens Wearers: Habitual comfilcon A Toric Lens Wearers
  Interventions: Device: comfilcon A Toric lens
- comfilcon A Multifocal Lens Wearers: Habitual comfilcon A Multifocal Lens Wearers
  Interventions: Device: comfilcon A Multifocal lens
- comfilcon A Multifocal Toric Lens Wearers: Habitual comfilcon A Multifocal Toric Lens Wearers
  Interventions: Device: comfilcon A Multifocal Toric lens
- comfilcon A Energys Lens Wearers: Habitual comfilcon A Energys Lens Wearers
  Interventions: Device: comfilcon A Energys lens

INTERVENTIONS:
Device: comfilcon A Sphere lens — 2 hours of wear
  Groups: comfilcon A Sphere Lens Wearers
Device: comfilcon A Toric lens — 2 hours of wear
  Groups: comfilcon A Toric Lens Wearers
Device: comfilcon A Multifocal lens — 2 hours of wear
  Groups: comfilcon A Multifocal Lens Wearers
Device: comfilcon A Multifocal Toric lens — 2 hours of wear
  Groups: comfilcon A Multifocal Toric Lens Wearers
Device: comfilcon A Energys lens — 2 hours of wear
  Groups: comfilcon A Energys Lens Wearers

SUMMARY:
The main objective of this study is to demonstrate acceptable safety and effectiveness (performance) of comfilcon A Sphere, Toric, Multifocal, Toric Multifocal and Energys lenses, when used in the general population.

DETAILED DESCRIPTION:
The main objective of this study is to demonstrate acceptable safety and effectiveness (performance) of comfilcon A Sphere, Toric, Multifocal, Toric Multifocal and Energys lenses, when used in the general population after 2 hours of wear.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 to 75 years (inclusive).
2. Current wearer of the Comfilcon A sphere, toric, multifocal, toric multifocal or Energys contact lens for at least 12 months.
3. At least occasional overnight wear in the last 12 months.

Exclusion Criteria:

1. Current participation in a contact lens or contact lens care product clinical trial.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female or male subjects aged 8 to 75 years who are established contact lens wearers. Screen and enrol approximately 182 participants wearing comfilcon A lenses with the aim of achieving at least 160 in the per protocol analysis cohort.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual Performance (Visual Acuity) | At the end of 2 hours of wear
  Visual Performance will be measured using logMAR
  * High contrast, high illumination distance VA
  * High contrast, high illumination near VA
Incidence of contact lens-related adverse events | At the end of 2 hours of wear
  Incidence of contact lens-related adverse events will be recorded from subjects

CONTACTS AND LOCATIONS:
Overall Officials: Meng C Lin, OD, PhD, Principal Investigator — University of Berkeley; Katherine Bickle, Dr., Principal Investigator — ProCare Vision Center; Abigail G Harsch, Dr., Principal Investigator — Nittany Eye Associates; David Browning, Dr., Principal Investigator — Drs. McIntyre, Garza, Avila and Jurica, Optometrists
Locations (4):
- United States (4):
  - University of Berkeley, Berkeley, California
  - ProCare Vision Center, Granville, Ohio
  - Nittany Eye Associates, College, Pennsylvania
  - Drs. McIntyre, Garza, Avila and Jurica, Optometrists, Corpus Christi, Texas